CLINICAL TRIAL: NCT00418756
Title: A Phase I Open-label, Two Period, Single Center Study to Assess the Effect of 600 mg Daily Oral Dose of Rifampin (CYP3A4 Inducer) on the Pharmacokinetics of a Single 400 mg Oral Dose of Nilotinib in Healthy Subjects
Brief Title: Effects of Rifampin on the Pharmacokinetics of Nilotinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2115
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: nilotinib; Rifampin; PK; healthy subjects
MeSH Terms: interventions — nilotinib

ARMS (1):
- Rifampin + nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Semi-synthetic antibiotic derivative of rifamycin B and is known to induce cytochrome P-450 (CYP) enzymes.
  Other Names: AMN107A, Tasigna

SUMMARY:
This study will evaluate the effect of 600 mg daily oral dose of rifampin (CYP3A4 inducer) on the pharmacokinetics of a single 400 mg oral dose of nilotinib in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male (18 - 55 yrs) and sterile or post menopausal female subjects:
2. Body weight must be ≥50 kg and <100 kg, with a body mass index (BMI) >18 but <33.

Exclusion Criteria:

1. Female who is pregnant, test positive for a serum pregnancy test or currently breast feeding.
2. Contraindication to receiving nilotinib or rifampin.
3. Smokers or use of tobacco products or products containing nicotine in the last 30 days
4. A past medical history of clinically significant Electrocardiogram abnormalities, or a history/family history of long QT-interval syndrome.

Other protocol-defined inclusion/exclusion may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of 600 mg rifampin on the pharmacokinetics (PK) of a single 400mg (2 x 200mg capsules) oral dose of AMN107 | at pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose after AMN107 administration on Days 1 and 16.

SECONDARY OUTCOMES:
To assess the safety and tolerability of a single 400mg (2x200mg capsules) oral dose of AMN107 given alone and concomitantly with 600mg rifampin
To determine the ratio of 6ß - hydroxylcortisol to cortisol in urine as an in-vivomarker of CYP3A4 induction with rifampin treatment4. | on Days -1, 11, 15 and 19

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals